CLINICAL TRIAL: NCT04006405
Title: AURORAX-0087A: Glycosaminoglycan Scores for Surveillance of Recurrence in Leibovich Points ≥5 Non-metastatic Clear Cell Renal Cell Carcinoma
Brief Title: AURORAX-0087A: GAG Scores for Surveillance of Recurrence in Leibovich Points ≥5 Non-metastatic ccRCC
Acronym: AUR87A
Status: Completed | Type: Observational
Sponsor: Elypta (Industry)
Responsible Party: Sponsor
Other Study IDs: ECD-AUR87A001
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: 140 patients with a minimum follow-up of 12 months
  Interventions: Diagnostic Test: GAG score
- Cohort 2: up to 140 patients with a minimum follow-up of 12 months
  Interventions: Diagnostic Test: GAG score

INTERVENTIONS:
Diagnostic Test: GAG score — blood and urine samples to determine GAG scores

SUMMARY:
AUR87A is an observational prospective multicenter diagnostics test cohort study for detection of renal cell carcinoma recurrence as determined by the reference standard, which is imaging using computed tomography (CT) of the chest and abdomen at defined intervals after primary surgery.

DETAILED DESCRIPTION:
Non-metastatic clear cell renal cell carcinoma (ccRCC) recur in ~20% of cases within 5 years after radical surgery. Current postoperative follow-up protocols, being schematic and at best based on risk of recurrence scores, are sub-optimal for early detection of recurrences which could potentially be available for curative management. Blood and urine collected glycosaminoglycans (GAGs) are promising novel class of biomarkers from which a new diagnostic test based on so called GAG scores has been developed. GAG scores have accurately distinguished localized/locally-advanced and advanced RCC from healthy subjects.

AUR87A features an adaptive design. The primary endpoint analysis is conducted when 30 events (i.e. recurrences) are reached - expected at 140 patients with a minimum follow-up of 12 months (cohort 1). An interim analysis at 15 events is conducted to verify whether the sensitivity and specificity estimates are in line with the study assumptions. In case of futility, the GAG scores formulations and/or cut-offs are optimized based on data from cohort 1. The primary endpoints are then validated on a second independent cohort, powered depending on the results from cohort 1. This second cohort is estimated in 140 patients (cohort 2). In case of non-futility, cohort 2 may be used as external validation.

AUR87A will prospectively enroll an estimated 280 non-metastatic ccRCC patients curatively treated with surgery (partial or radical nephrectomy). Patients are followed-up longitudinally using GAG scores in blood and urine every 3 months after surgery, alongside the current standard follow-up protocol, i.e. imaging, as reference standard.

The hypothesis of AUR87A is that postoperative increase of the GAG scores, so called "GAG recurrence ", can predict or detect recurrence at an earlier time-point compared to the reference standard, referred to as "radiological recurrence", and thereby improve the clinical utility of current follow-up protocols.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening inclusion criteria

* Size of primary tumor >4cm (>cT1a) in greatest dimension on pre-operative abdominal CT-scan
* Size of primary tumor ≤4cm is allowed if pre-operative abdominal CT-scan shows suspected RCCs with radiological sign of venous tumor thrombus (renal vein or caval).
* Pre-operative CT-scan of chest and abdomen show no signs of metastatic disease
* Localized and biopsy proven clear cell RCC (ccRCC) under active surveillance which at timepoint of study recruitment, opted for surgery because of growth rate of primary tumor to a size > 4cm
* Elected for curative intent surgery for RCC

Final screening inclusion criteria

* Any gender being 18 years or older at timepoint of final inclusion
* In postoperative pathology report shown to be ccRCC subtype according to 8th Edition of the American Joint Committee on Cancer (AJCC)
* Leibovich points (LP) ≥5 according to Leibovich score system (2003)
* If pathology report shows multiple subtypes in same tumor, as long as the majority of tumor is ccRCC (>50%), participant can be included

Exclusion Criteria:

Pre-screening exclusion criteria

* TNM-stage T(any) N(any) M1 according to AJCC, i.e. metastatic disease at diagnosis
* Absence of preoperative chest imaging (chest CT) within 60 days prior to primary surgery
* Previous history of curatively treated for other cancers, still not deemed fully cured and participant still under surveillance for said cancer
* Participants offered active surveillance for RCC instead of curative intent surgery
* Participants offered any type of thermal ablation treatment instead of surgery, i.e. LP cannot be assessed

Final screening exclusion criteria

* Participants with AJCC cN0 status at preoperative imaging in whom a clinically suspicious regional lymph-node metastases (enlarged lymph node(s)) is noted during primary surgery, but who subsequently do not undergo any lymph node dissection. (Note: participants with cN0 status at pre-operative imaging and no clinical signs of regional lymph node metastases during primary surgery can still be included irrespective of lymph node dissection having been performed, i.e. being pN0 or pN1 if it is performed or pNx if it is not performed)
* Participants with AJCC cN1 status at pre-operative imaging in which lymph node dissection is not performed (i.e. pNx).
* Elected for any adjuvant therapy (i.e. systemic therapy) outside or within any clinical study
* Non-clear cell RCC histology or benign tumor (i.e. oncocytoma and angiomyolipoma, which are the most common benign types, but also any other rare types of benign renal tumors) after pathological analysis
* Any hereditary form of RCC (e.g. Von Hippel-Lindau, Birt-Hogg-Dubé, Hereditary Papillary RCC)
* RCC with pure sarcomatoid differentiation, also called sarcoma of the kidney
* Previous history of curatively treated for RCC with a suspected de novo RCC in the remaining kidney tissue
* Prior or current use of instillation therapy with hyaluronic acid and/or chondroitin sulfate (HA-CS).
* Use of heparin, including low molecular weight heparin (e.g. Enoxaparin, Dalteparin, Tinzaparin) for concurrent disease in need of blood dilution (e.g. ongoing deep vein thrombosis or lung emboli). Note: use of of heparin for thrombus prophylaxis in conjunction with primary surgery or postoperatively ≤4 weeks will be allowed.
* Patients who were not radically operated during primary surgery with the exception of histological positive surgical margin in participants who have undergone partial nephrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is a representative sample of the North American and European population of ccRCC patients with LP ≥ 5 after curative intent surgery
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of GAG recurrence | minimum follow-up of 12 months
  Sensitivity and specificity of GAG recurrence to LP≥5 ccRCC radiological or histologically verified recurrence with a minimum follow-up time of 12 months

SECONDARY OUTCOMES:
Absolute and relative risk increase (ARI/RRI) of radiological recurrence | within 6 months since last GAG score evaluation
  Absolute and relative risk increase (ARI/RRI) of radiological recurrence in patients with GAG recurrence versus no GAG recurrence
Recurrence-free survival (RFS) | minimum follow-up of 12 months
  Recurrence-free survival (RFS) in the LP≥5 ccRCC for GAG recurrence vs. no GAG recurrence with a minimum follow-up time of 12 months
Positive and negative predictive value (PPV/NPV) of GAG recurrence | minimum follow-up of 12 months
  Positive and negative predictive value (PPV/NPV) of GAG recurrence to LP ≥5 ccRCC radiological recurrence
Area under the receiver-operating-characteristic curve (AUC) of GAG scores | minimum follow-up of 12 months
  Area under the receiver-operating-characteristic curve (AUC) of GAG scores to LP ≥5 ccRCC radiological recurrence
RFS, overall survival (OS) and cancer specific survival (CSS) | follow-up time of 2 years and 5 years respectively after primary surgery
  RFS, overall survival (OS) and cancer specific survival (CSS) in patients with GAG recurrence versus no GAG recurrence
Concordance-index (C-index) of preoperative GAG scores | follow-up time of 2 years and 5 years respectively after primary surgery
  Concordance-index (C-index) of preoperative GAG scores versus risk nomograms for RFS and for CSS
Lead-time GAG vs. radiological recurrence among true positives | minimum follow-up of 12 months
  Lead-time GAG vs. radiological recurrence among true positives

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Dabestani, Principal Investigator — Lund University, Dept. Clinical Sciences, Skåne University Hospital
Locations (29):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- UZ Leuven, Leuven, Belgium
- Prostate Cancer Centre, Calgary, Canada
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- Helsinki University Central Hospital, Helsinki, Finland
- Hôpital Henri Mondor, Créteil, France
- Italy (6):
  - AOU San Orsola Malpighi, Bologna
  - Careggi University Hospital, Florence
  - San Raffaele Hospital, Milan
  - AOU San Luigi Gonzaga, Orbassano
  - Istituto Nazionale Tumori Regina Elena, Roma
  - AOU Integrata Verona, Verona
- Hospital da Luz Coimbra, Coimbra, Portugal
- Spain (2):
  - Hospital Universitario Cabueñes, Gijón
  - University Hospital of Valencia, Valencia
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Norrlands University Hospital, Umeå
- United Kingdom (8):
  - Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Frimley Park Hospital, Frimley
  - Guys & St Thomas Hospital, London
  - Royal Free Hospital, London
  - Norfolk & Norwich University Hospital, Norwich
  - Royal Berkshire Hospital, Reading
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified clinical and biochemical data will become available to the research community along with the publication of a scientific article related to the present investigation.

REFERENCES:
- See also: Official website for AURORAX-87A — https://elypta.com